CLINICAL TRIAL: NCT03222518
Title: NSAIDs Versus Paracetamol Versus Paracetamol + NSAIDs in Traumatic Pain Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAR vs NSAIDs vs Comb in Pain
Record Dates: First submitted 2017-05-14; First posted 2017-07-19 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Acute Pain Due to Trauma
Keywords: acute pain, trauma, paracetamol, NSAID
MeSH Terms: conditions — Acute Pain; Wounds and Injuries | interventions — Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal; Piroxicam

STUDY DESIGN:
Intervention Model Description: Subjects are randomized in 3 arms:
  * paracetamol group
  * NSAID group
  * paracetamol + NSAID group
Who Masked: Participant, Outcomes Assessor
Masking Description: study medications consists of identical shape pills of each study medication randomization is made by sealed envelops and a randomly sequence generated numbers.
  patients and the research associate who collected the outcome data are blinded from the study group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Parcetamol Group (Active Comparator): The patient receives an envelope containing Paracetamol 1000 mg at the dose of 3 times / day + follow-up sheet + appointment card.
  Interventions: Drug: NSAID; Drug: paracetamol-NSAID
- NSAID Group (Active Comparator): The patient receives an envelope containing NSAID 20 mg piroxicam twice daily / day + follow-up sheet + appointment card.
  Interventions: Drug: Paracetamol; Drug: paracetamol-NSAID
- NSAID + Paracetamol Group (Active Comparator): The patient receives an envelope containing NSAID 20 mg piroxicam at a dose of 2 times/day + Paracetamol 1000 mg at a dose of 3 times / day + follow-up sheet + appointment card.
  Interventions: Drug: Paracetamol; Drug: NSAID

INTERVENTIONS:
Drug: Paracetamol — 21 pills of Paracetamol 1000mg are provided with a preconised dose of 1 pill 3 times per day over 7 days period
  Arms: NSAID + Paracetamol Group; NSAID Group
Drug: NSAID — 14 pills of piroxicam 20 mg are provided with a preconised dose of 1 pill 2times per day over 7 days period
  Other Names: piroxicam
  Arms: NSAID + Paracetamol Group; Parcetamol Group
Drug: paracetamol-NSAID — 21 identical pills of paracetamol ith a preconised dose of 1 pill 3 times per day over 7 days period+14 pills of piroxicam 20 mg are provided with a preconised dose of 1 pill 2times per day over 7 days period
  Other Names: combination
  Arms: NSAID Group; Parcetamol Group

SUMMARY:
The purpose of this study is to:

Compare the effect of paracetamol alone against NSAIDs alone against the association of paracetamol + NSAIDs in the treatment of traumatic pain.

DETAILED DESCRIPTION:
Paracetamol, NSAIDs, or a combination of the two molecules are usually prescribed. Patients even use these medications without a prescription. It is not known, however, whether or not NSAIDs have an additional value relative to paracetamol for the treatment of pain.

All patients were assigned in a 1:1:1 ratio. Randomization of subjects was performed centrally according to a computer-generated random code provided by one of investigators who was not involved in any other part of the trial. The patients included were divided into 3 groups: Paracetamol group who received paracetamol 1000 mg orally every 8th hour for 7 days; NSAID group who received piroxicam 20 mg orally twice a day for 7 days, and Paracetamol-NSAID combination who received both treatments at the same doses for 7 days. All protocol treatments were administered in opaque packets with code number according to the randomization list by an independent nurse who was not involved in monitoring or follow-up of the individuals. Data were collected for each patient, including demographics, medical history, and findings of the clinical examination. Injury Severity Score (ISS) whose values range from 0 to 75 was also assessed. Each patient was re-evaluated on the 3rd and 7th day post-trauma (D7) using a telephone contact by a clinical research associates who was blinded to the details of the study to note the following clinical data: pain VNS, ED readmissions for residual pain, need for other analgesics other than those of the protocol, other treatment modalities the patient might have used (adherence to the treatment prescribed), and side effects. In addition patients were asked about their satisfaction with pain control following ED using five point Likert scale: very dissatisfied, not satisfied, neutral, satisfied and very satisfied and about the degree to which they adhered to medication schedule. The principal investigator who was aware of the allocation was not involved in monitoring or recording of the outcomes until the data collection was completed.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* acute (<24 hours) post traumatic pain of the extremity and requiring analgesic treatment upon discharge for pain with intensity >3 on a visual numeric scale

Exclusion criteria:

* open fracture
* head, abdominal, thoracic or polytrauma.
* Need for hospitalization, regular use of paracetamol and NSAIDs during the two weeks before admission to ED
* history of allergy or hypersensitivity to either paracetamol or NSAIDs,
* contraindication to paracetamol or NSAIDs,
* acute /history of GI hemorrhage and renal insufficiency,
* an inability to assess pain intensity according to the VNS.
* Pregnancy
* heart failure
* known hepatic cirrhosis
* known severe renal impairment (Creatinine clearance <30 ml/min)
* swallowing disorders
* Refusal, incapacity or difficulties to consent or to communicate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
new oral analgesic medications needed rate | 3 days and 7 days
  oral analgesic medications other than those of the protocol prescribed by the treating physicians or taken by patients' own volition

SECONDARY OUTCOMES:
the between-group difference in mean change in VNS score measured from ED discharge (VNS D0) to 7 days later | 3 and 7 days
  [delta VNS= (VNS D0 - VNS D7 / VNS D0) x 100]
The appearance of side effects | 7 days
  The appearance of side effects: such as Drowsiness ,Decreased respiratory rate (<14 c / min), Cutaneous rash, Vomiting,Nausea,pruritus, Dizziness.
  • Digestive hemorrhage.
the rate of ED readmissions for residual pain | 3 and 7 days
  ED readmissions for residual pain
patient satisfaction assessed by Likert's verbal scale. | 3 and 7 days
  patient satisfaction assessed by Likert's verbal scale.

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, MD, Principal Investigator — University of Monastir
Locations (1):
- Monastir University Hospital, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No